CLINICAL TRIAL: NCT03053765
Title: Optimizing Fidelity of Interpersonal Psychotherapy for Depression
Brief Title: Optimizing Fidelity of Interpersonal Psychotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Conflict of Interest (COI) cannot be managed
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R33MH097041 (NIH)
Record Dates: First submitted 2016-08-09; First posted 2017-02-15 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Individual Supervision in IPT (Active Comparator): Bi-weekly individual case supervision in IPT
  Interventions: Other: training in IPT
- Group Supervision in IPT (Experimental): Bi-weekly group supervision in IPT in groups of 4-6 therapists
  Interventions: Other: training in IPT
- Internet-Based Training in IPT (Experimental): Access to internet-based training in IPT to review information learned in initial 2-day training
  Interventions: Other: training in IPT
- Autodidactic Training in IPT (No Intervention): Clinicians allowed access to training materials and can engage in self-study

INTERVENTIONS:
Other: training in IPT — Follow-up training in IPT to determine which best enhances fidelity
  Arms: Group Supervision in IPT; Individual Supervision in IPT; Internet-Based Training in IPT

SUMMARY:
The study is designed to develop and validate an instrument to measure quality and adherence to IPT for research and training purposes. The measure is now being used to evaluate training in IPT.

DETAILED DESCRIPTION:
The study is a randomized trial comparing 4 different methods of follow-up training in IPT. Following initial 2-day training, participant therapists will be randomized to either individual supervision, group supervision, an internet-based training program, or autodidactic training. Participants will be followed for a year to determine their use of IPT, outcomes with patients, and adherence and quality of IPT in 4 case portfolios. The adherence measure for IPT developed in Phase I of the project is being used as the gold standard measure of IPT fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Active and licensed therapist conducting psychotherapy treatment; naïve to training in IPT

Exclusion Criteria:

* Inactive or not treating patients

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-08-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
expert evaluation of conduct of IPT using IPT Quality and Adherence Measure | one year
  The "IPT Quality and Adherence Measure" is the title of a single outcome measure used to assess clinicians performance of IPT

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stuart, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States